CLINICAL TRIAL: NCT05249556
Title: Double-blind, Randomized, Placebo-controlled Trial of Adjunctive Ganaxolone in the Treatment of Seizures Associated With Genetically Confirmed Cyclin-dependent Kinase-like 5 (CDKL5) Deficiency Disorder (CDD) in Pediatric Patients From 6 Months to Less Than 2 Years of Age.
Brief Title: Double-blind, Randomized, Placebo-controlled Trial of Ganaxolone in CDKL5 Deficiency Patients 6 Months to Less Than 2 Years Old
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immedica Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1042-CDD-3002
Record Dates: First submitted 2022-01-27; First posted 2022-02-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: CDKL5 Deficiency Disorder
MeSH Terms: conditions — CDKL5 deficiency disorder | interventions — ganaxolone; Bulk Drugs

STUDY DESIGN:
Intervention Model Description: This is a global, double-blind, randomized, PBO-controlled trial of adjunctive GNX treatment in participants 6 months to less than 2 years of age with genetically confirmed CDD
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator and research staff will be aware of the ascending dose design of the clinical investigation; however, the investigator, the research staff, and the participants will be blinded with respect to who is receiving active drug versus PBO.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GNX (Experimental): The suspension contains GNX (50 mg/mL), hydroxypropyl methylcellulose, polyvinyl alcohol, sodium lauryl sulfate, simethicone, methylparaben, propylparaben, citric acid, and sodium citrate at pH 3.5 to 4.2, and is sweetened with sucralose and flavored with artificial cherry.
  Interventions: Drug: Ganaxolone
- Placebo (Placebo Comparator): The PBO suspension consists of titanium dioxide, Avicel® (microcrystalline cellulose and carboxymethylcellulose sodium), sodium lauryl sulfate, simethicone, methylparaben, propylparaben, citric acid, sodium citrate and is sweetened with sucralose and flavored with artificial cherry
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ganaxolone — Ganaxolone
  Other Names: Active Drug
  Arms: GNX
Drug: Placebo — Placebo (for ganaxolone)
  Other Names: Inactive
  Arms: Placebo

SUMMARY:
This study will assess the efficacy, safety, and tolerability of ganaxolone (GNX) compared with placebo (PBO) as adjunctive therapy to the participant's standard anti-epileptic medication for the treatment of seizures in pediatric patients from 6 months to less than 2 years old with genetically confirmed CDD during a 12-week, DB phase. Pharmacokinetic (PK) assessments and population PK analyses will also be performed during this time. The DB phase will be followed by an optional long-term OL phase at which time all participants will receive GNX as an adjunct to their standard anti-seizure medication. Efficacy, safety and tolerability, and PK assessments will continue to be performed.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of CDD, including molecular confirmation of a pathogenic or likely pathogenic CDKL5 variant and refractory seizures (see Inclusion criterion 5).

   1. The principal investigator (PI) must review the results of the genetic analysis and confirm that gene mutation is likely to be the cause of the epilepsy syndrome.
   2. If the participant has a de novo variant of unknown significance (VUS) in the kinase domain of the CDKL5 gene, parental testing is negative and meets all other inclusion criteria, then the participant can be included.
   3. Genetic mutations will be confirmed by the sponsor's chosen central laboratory. In France, genetic mutations may be confirmed by an approved French organization, in compliance with French legislation prior to Screening/Visit 1.
2. Male or female participants aged 6 months to less than 2 years.
3. Parent(s) or LAR willing to give written informed consent, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures.
4. Failure to control seizures despite appropriate trial of 1 or more anti-seizure medications at therapeutic doses.
5. Have a history of at least 8 countable seizures during the 28 days prior to screening. Countable seizures will be defined by the following:

   1. Seizures with or without impairment of consciousness with a clear motor component, including generalized tonic-clonic, focal to bilateral tonic-clonic, atonic, bilateral clonic, bilateral tonic, focal motor seizures with or without impaired awareness, or infantile spasms. Clusters of infantile spasms/tonic seizures will be counted as a single seizure.
   2. Excludes myoclonic, absence or focal aware seizures without a clear motor component.
6. Participants should be on a stable regimen of anti-seizure medications for ≥ 2 weeks prior to the screening visit, without a foreseeable change in dosing for the duration of the DB phase.

   1. Concurrent use of adrenocorticotropic hormone (ACTH), prednisone or other glucocorticoids or vigabatrin are permitted.
   2. Vagus nerve stimulator (VNS) settings, ketogenic diet, or a modified Atkins diet should be unchanged for 1 month prior to screening and throughout the study (until the end of the DB phase).
7. Use of dietary supplements or herbal preparations is permitted if the participant has been using them consistently for more than 1 month prior to screening and there is no plan on changing the dose for the duration of the DB phase.
8. Parent/caregiver is able and willing to maintain an accurate and complete daily seizure eDiary for the duration of the study.
9. Able and willing to administer IP with food 3 times daily.

Exclusion Criteria:

1. Have an active CNS infection, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive as evaluated by brain imaging (magnetic resonance imaging [MRI]).
2. Have any disease or condition (medical or surgical; other than CDKL5 deficiency) at screening that might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or hepatic systems; or other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the IP, or would place the participant at increased risk.
3. Has a positive result for tetrahydrocannabinol (THC) test (via urine or plasma drug screen) at the screening visit. Concomitant Epidiolex/Epidyolex (cannabidiol derivative [CBD]) use will be allowed in the DB phase provided the participant has been on a stable dose for at least 1 month prior to screening and is expected to remain on a stable dose without a foreseeable change for the duration of the DB phase.
4. Use of a CBD preparation other than Epidiolex/Epidyolex for 1 month prior to screening.
5. An AST (aspartate aminotransferase/serum glutamic-oxaloacetic transaminase [SGOT]) or ALT (alanine aminotransferase/serum glutamic-pyruvic transaminase [SGPT]) > 3 times the upper limit of normal (ULN) at study entry. If AST or ALT increases > 3 X ULN during the study, the participant should be followed with weekly laboratory repeat testing and continue in study if levels trending down. The participant will be discontinued if levels do not decline to < 3 X ULN.
6. Total bilirubin levels greater than the ULN at study entry. In cases of a documented, stable medical condition (ie, Gilbert's Syndrome) resulting in levels of total bilirubin greater than the ULN, the medical monitor can determine if a protocol exception can be made. If total bilirubin increases to 1.5 x the ULN or more during study, the participant will be discontinued.
7. Participants with significant renal insufficiency, with an estimated glomerular filtration rate (eGFR) < 30 mL/min (calculated using the Cockcroft-Gault formula or Pediatric GFR calculator or Bedside Schwartz).
8. Using St. John's Wort.
9. Have been exposed to any other investigational drug within 30 days or less than 5 half-lives prior to screening.
10. Known allergic reaction or sensitivity to GNX or its excipients.
11. Participating in any other study involving administration of an investigational medication or device.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Percent Change from baseline in 28-day frequency of countable seizures | Baseline through 12 weeks
  Percent change from baseline in 28-day frequency of countable seizures through the end of the 12-week, DB treatment phase relative to the 4-week prospective baseline phase

SECONDARY OUTCOMES:
Percentage of participants experiencing >50% reduction | Baseline through 12-week DB phase
  Percentage of participants experiencing ≥ 50% reduction in the 28-day primary frequency of all countable seizures compared to a 4-week baseline
Percent change from baseline in 28-day frequency of countable seizures through maintenance phase | Baseline through Double-Blind & Maintenance
  Percent change from baseline in 28-day frequency of countable seizures during the Maintenance Period of the DB phase
Percent change in seizures by seizure type | Baseline through 12-week DB phase
  Percent change in seizures by seizure type
Percent change in seizure-free days | Baseline through 12-week DB phase
  Percent change in seizure-free days
CGI-I at the end of the 12-week DB phase | Baseline through 12-week DB phase
  CGI-I (Caregiver Global Impression of Improvement) at the end of the 12-week DB phase (further details to be described)
CGI-CSID at the end of the 12-week DB phase | Baseline through 12-week DB phase
  CGI-CSID (Seizure Intensity/Duration) at the end of the 12-week DB phase

REFERENCES:
- [Derived] Yasmen N, Sluter MN, Yu Y, Jiang J. Ganaxolone for management of seizures associated with CDKL5 deficiency disorder. Trends Pharmacol Sci. 2023 Feb;44(2):128-129. doi: 10.1016/j.tips.2022.11.007. Epub 2022 Dec 12. No abstract available. PMID 36517284